CLINICAL TRIAL: NCT04269187
Title: Diaphragmatic Ultrasound in Critically Ill Patients With Therapeutic Theophylline Trials
Brief Title: Diaphragmatic Ultrasound With Theophylline Therapeutic Trials
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Roshdy Abdul Satar Mohamed, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUS in critically ill patients
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Diaphragmatic Dysfunction in Critically Ill Patients
MeSH Terms: interventions — Theophylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With theophylline treatment (Experimental): This group will be for: diaphragmatic ultrasound after admission to ICU and before administration of theophylline; 200 mg/d orally for 12 days then reassessment of diaphragm by ultrasound.
  Interventions: Drug: Theophylline
- No theophylline treatment (No Intervention): This group will be for: diaphragmatic ultrasound after admission to ICU then reassessment of diaphragm by ultrasound before discharge

INTERVENTIONS:
Drug: Theophylline — Theophylline oral 200 mg daily for 12 days
  Arms: With theophylline treatment

SUMMARY:
Critically ill patients are a group of patients with special needs during hospitalization. The vast majority of them is mechanically ventilated and requires continuous assessment of vital parameters.

It is quite impressive that assessment of respiratory muscles, and specifically of the diaphragm, is lacking in the daily practice of ICU.

The diaphragm-the main inspiratory muscle-is considered so important in ICU. A lot of time in ICUs is spent on weaning patients from mechanical ventilation. Although weaning from mechanical ventilation can be a rapid and uneventful process for the majority of the patients, it can be difficult in as many as 20-30% of them (1)(2). It is during weaning that the diaphragm becomes the major pathophysiological determinant of weaning failure or success.

Weaning failure is defined as failing a spontaneous breathing trial or developing a post-extubation respiratory distress that requires re-intubation or non-invasive ventilation within 48 h following extubation (3).

So, identification of reliable predictors of weaning failure may represent potential avenues of treatment that could reduce the incidence of weaning failure and its associated morbidity.

Known predictors of weaning failure include chronic obstructive airway disease (3), cardiac failure(4-6), lung de-recruitment (7), pneumonia (8) and diaphragmatic dysfunction (9).

Rapid shallow breathing index (RSBI) is a clinical predictor of failure of weaning from mechanical ventilation and it is widely used in clinical research and in practice (10).

However, diaphragmatic ultrasonography could be a promising tool for predicting reintubation within 48 hours of extubation. As it permits direct assessment of diaphragm function.

It should be mentioned that diaphragmatic dysfunction among patients hospitalized in the intensive care unit (ICU) is commonly attributed to critical illness polyneuropathy and myopathy. Mechanical ventilation, even after a short period of time, can also induce diaphragmatic dysfunction.

Recent researches have shown that theophylline improves diaphragmatic contractility in isolated muscle preparations in animals and in normal human subjects. The question now does the theophylline have a significant role in critical ill patients with diaphragmatic dysfunction whether they are diabetic or not ?

DETAILED DESCRIPTION:
All patients will be subjected to:

1. medical history.
2. clinical examination.
3. diaphragmatic ultrasound : diaphragmatic thickness and excursion will be assessed.
4. theophyllin treatment; 200 mg/d orally for 12 days then reassessment of diaphragm by ultrasound.
5. weaning trial ; Patients are considered ready for weaning when they meet all the following criteria: fraction of inspired oxygen (FiO2) < 0.5, positive end expiratory pressure (PEEP) ≤ 5 cm water , Pa O2/Fi O2> 200, respiratory rate (RR) <30 breaths/min, alert and cooperative, and hemodynamically stable in the absence of any vasopressor therapy support.(11)

   1. rapid shallow breathing index (RSBI) will be measured. It's defined as the ratio between the respiratory rate (breaths/min) and tidal volume (TV) (liters).
   2. 2-hour spontaneous breathing trial with a T-piece and zero pressure support (before extubation).
   3. extubation is done & follow up for 48 hours

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are as follows: critical ill patients that are admitted to our ICU whether they are mechanically ventilated or not .

Exclusion Criteria:

* exclusion criteria are the presence of pneumothorax or ascites, a history of either neuromuscular disease or thoracic surgery, congenital diaphragmatic hernia, the presence of a tracheostomy tube,chronic obstructive pulmonary disease (COPD) patients, asthma and poor image quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
how much improvement in diaphragmatic thickness and excursion after theophylline treatment. | Baseline
  how much improvement in diaphragmatic thickness and excursion after theophylline treatment.

SECONDARY OUTCOMES:
number of successful weaning trials based on diaphragmatic ultrasound findings | Baseline
  number of successful weaning trials based on diaphragmatic ultrasound findings

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Sharaf ElDin, Lecturer, Study Director — Assiut university; internal medicine department; Sahar Farghaly, Lecturer, Study Director — Assuit university; chest diseases department; Hanan Mahmoud, Professor, Study Director — Assuit university; internal medicine department

REFERENCES:
- [Background] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.
- [Background] Farghaly S, Hasan AA. Diaphragm ultrasound as a new method to predict extubation outcome in mechanically ventilated patients. Aust Crit Care. 2017 Jan;30(1):37-43. doi: 10.1016/j.aucc.2016.03.004. Epub 2016 Apr 22. PMID 27112953
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/7921460/
- See also: Related Info — https://www.google.com/url?sa=t&source=web&rct=j&url=https://daneshyari.com/article/preview/5562965.pdf&ved=2ahUKEwitvd-7m73nAhWmRhUIHX_jCRQQFjAAegQIAxAB&usg=AOvVaw3dzzyX2YgXmojGd_nnAw97